CLINICAL TRIAL: NCT03487887
Title: Continuous Glucose Monitoring in Patients With Diabetes Mellitus Type 2 in Secondary Care
Brief Title: Secondary Care - Continuous Glucose Monitoring
Acronym: SC-COSMO
Status: Completed | Type: Observational
Sponsor: Croatian Society for Endocrinology and Diabology (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Maja Baretić, Principal investigator Maja Baretić MD PhD, Croatian Society for Endocrinology and Diabology
Other Study IDs: Program CGM u bolesnika T2DM
Record Dates: First submitted 2018-03-21; First posted 2018-04-04 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: continuous glucose monitoring; glycemic variability; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: continuous glucose monitoring (CGM) iPro™2 Medtronic — A CGM device is to be set and take off by the diabetologist. Before the study start all diabetologist not familiar to the method will have a short education on CGM device. Study period is seven days and includes screening before study entry and two visits. On Day 1, after screening and signing the informed consent, the CGM device is applied. Patient is instructed to keep a 7 day diary with four daily standard SMBG along with the data on eating, physical exercise, drugs. On Day 7, CGM device is taken off and the data from iPro2 is uploaded to PC. At the end, each patient fills a short query on satisfaction while wearing CGM.

SUMMARY:
Introduction and objective: The current state of glucose monitoring includes the use of A1C, self-monitoring of blood glucose (SMBG), and continuous glucose monitoring (CGM). CGM technology has got the potential to revolutionize diabetes care in the near future striving to optimal diabetes management and tight glucose control. Until very recently, this determination could only be achieved by the attainment of multiple capillary blood glucose determinations each day and/or measuring hemoglobin A1C. Those methods are not accurate in cases of unrecognized hypoglycemia, unrecognized nighttime events or in cases of large swings in blood glucose. Our aim is to analyze the benefit of tracking patterns of glucose values by using professional CGM technology used for "blinded" collection of glucose data retrospectively in patients with T2DM in secondary care- diabetologist clinic.

DETAILED DESCRIPTION:
STUDY DESIGN: An observational, multicenter, cross-sectional study. A total of 20 diabetologist from four Croatian regions will recruit up to ten subjects of both sexes from May 2018 till the end of May 2019, diagnosed with type 2 diabetes mellitus at least one year prior to study entry, aged ≥40 years, with only basal insulin in therapy and with clinical suspicion of hypoglycemia or with disproportion in actual glycaemia and hemoglobin A1c findings. Sociodemographic, laboratory (HbA1c, fasting and postprandial glucose, total cholesterol, and high density cholesterol, and low density cholesterol, triglyceride and serum creatinine) and habits data will be collected.

SETTING: Totally 100 of patients will be included. At diabetologist office each patient wear the device (iPro™2 Medtronic) subcutaneously for up to 7-days and return it to the office for download. Patients only see the CGM data after it's been analyzed by the healthcare professional. A CGM device is to be set and take off by the diabetologist. Before the study start all diabetologist who are not familiar to the method will have a short education. Study period is seven days and includes screening before study entry and two visits. On Day 1, after screening and signing the informed consent, the CGM device is applied. Patient is instructed to keep a 7 day diary with four daily standard SMBG along with the data on eating, physical exercise, drugs. On Day 7, CGM device is taken off and the data from iPro2 is uploaded to PC. At the end, each patient fills a short query on satisfaction while wearing CGM.

ELIGIBILITY:
Inclusion Criteria:

* T2DM diagnosed at least one year prior to study entry
* Only basal insulin in therapy
* Patients' ability to understand and answer the questionnaire by themselves
* Signed informed consent

Exclusion Criteria:

* Known coagulopathy
* Oral anticoagulants in therapy
* Skin disease that enables continuous glucose monitor device application
* Febrile illness
* Patient's inability to physically visit a general practitioners office
* Patient's inability to answer the questionnaire by themselves

Ages: 3 Days to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Totally 100 of patients with type 2 diabetes mellitus diagnosed at least one year prior to study entry, aged ≥40 years, both sexes, treated in secondary care, with no insulin in therapy and with clinical suspicion of hypoglycemia or with disproportion in actual glycaemia and A1C findings will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Glycemic variability | 7 days
  Glycemic variability measured by continuous glucose monitor devicein individuals with type 2 diabetes mellitus in secondary care

SECONDARY OUTCOMES:
Hypogliaemia | 7 days
  Hypogliaemia measured by continuous glucose monitor device in individuals with type 2 diabetes mellitus in secondary care

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No